CLINICAL TRIAL: NCT00504296
Title: A Phase I Clinical and Pharmacokinetic Study of SB939 in Patients With Advanced Cancer
Brief Title: SB939 in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: S*BIO (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I188; CAN-NCIC-IND188 (Registry Identifier: NCI US - Physician Data Query); S*BIO-SB939-2007-002 (Other: S*BIO); CDR0000558934 (Other: PDQ)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — SB939 compound; Immunoenzyme Techniques; Immunohistochemistry; Immunologic Techniques; Chromatography, Liquid; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SB939 (Experimental)
  Interventions: Drug: HDAC inhibitor SB939; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: immunologic technique; Other: laboratory biomarker analysis; Other: liquid chromatography; Other: mass spectrometry; Other: pharmacological study

INTERVENTIONS:
Drug: HDAC inhibitor SB939 — SB939 will be administered initially for 3 consecutive days every other week at the first dose level and then for 5 consecutive days every other week at escalating doses.
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: immunologic technique
Other: laboratory biomarker analysis
Other: liquid chromatography
Other: mass spectrometry
Other: pharmacological study

SUMMARY:
RATIONALE: SB939 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of SB939 in treating patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the recommended phase II dose of oral SB939 in patients with solid tumors.

Secondary

* To determine the toxic effects of SB939 and its association with dose and pharmacokinetics.
* To assess the pharmacokinetic profile of SB939.
* To assess preliminary evidence of antitumor effects of SB939 in patients with measurable disease as documented by objective response.
* To establish proof-of-principle for SB939 effects on histone acetylation by evaluation of histone acetylation and other biomarkers in peripheral blood mononuclear cells (PBMCs) at all dose levels.

OUTLINE: Patients receive oral SB939 once daily on days 1-5 and 15-19. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically during course 1 for pharmacokinetic and pharmacodynamic studies. Samples are analyzed for levels of SB939 via LC-MS/MS method and levels of acetylated histone 3 (AcH3), target effect, downstream consequences, and tumor response via western blot, immunohistochemistry, or ELISA methods.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumor

  * Refractory to standard therapy or for which conventional therapy is not reliably effective

Exclusion criteria:

* Patients with documented CNS metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status of 0, 1, or 2
* Must have a life expectancy of ≥ 12 weeks
* Granulocytes (AGC) ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Bilirubin ≤ upper limit of normal (ULN)
* AST and ALT ≤ 2.5 x ULN (< 5 x ULN if liver metastases are present)
* Serum creatinine ≤ 1.2 x ULN OR creatinine clearance ≥ 60 mL/min
* QTc ≤ 450 msec
* LVEF ≥ 50% by ECHO or MUGA
* Troponin I or T ≤ ULN
* Must be within 1½ hour's driving distance

Exclusion criteria:

* Pathologic cardiac arrhythmia requiring active treatment

  * Patients with a history of arrhythmia must be > 12 months since last treatment with no recurrence of arrhythmia in the interval
* Inability to take oral medication

  * Patients must be able to swallow SB939 capsules and have no gastrointestinal abnormalities (e.g., bowel obstruction or previous gastric resection) which would lead to inadequate absorption of SB939
* Pregnant or lactating women

  * Urine or serum B-HCG must be negative
* Women or men of child-bearing potential unless using effective contraception
* Presence of any clinically significant co-morbidities (i.e., pulmonary disease, active CNS disease, or active infection)
* Presence of any other significant CNS disorder that would hamper the patient's compliance
* Presence of any significant psychiatric disorder that would hamper the patient's compliance
* Other acute or chronic medical condition, psychiatric condition, or laboratory abnormality that may increase the risks associated with study participation/study drug administration or may interfere with the interpretation of study results
* Pre-existing peripheral neuropathy ≥ grade 2
* Known HIV or hepatitis B or C infection

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Previous anticancer treatment must be discontinued at least 28 days prior to the first dose of study treatment (42 days [6 weeks] for nitrosoureas or mitomycin C)
* At least 28 days since prior radiation therapy restricted to ≤ 30% of the bone marrow and recovered from toxic effects

  * Exceptions may be made for low-dose nonmyelosuppressive radiotherapy
* Must be ≥ 14 days since any major surgery
* Pre-existing bisphosphonate or luteinizing hormone-releasing hormone (LHRH) analog therapy (for men with hormone refractory prostate cancer) may be continued during study participation

Exclusion criteria:

* Previous treatment with a histone deacetylase (HDAC) inhibitor
* Treatment with another investigational therapy within 28 days prior to study entry
* Other concurrent anticancer treatment or investigational therapy
* Concurrent agents with a known risk of Torsade de Pointes
* Concurrent G-CSF, GM-CSF, or other hematopoietic growth factors may not be used as a substitute for a scheduled dose reduction (may be used in the management of acute toxicity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-09-14 (Actual); Primary Completion 2010-04-22 (Actual); Study Completion 2011-06-21 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose | Each dose level
  Assess for safety, tolerability, toxicity profile and dose limiting toxicities

SECONDARY OUTCOMES:
Safety | Each dose level
  Safety, tolerability, toxicity profile, dose limiting toxicities of SB939.
Pharmacokinetic profile | Cycle 1 day 1 and 15
  Samples collected over multiple timepoints
SB939 effects on histone H3 acetylation | Cycle 1 days 1 and 15
  Levels of AcH3 will be determined using wetern Blot, immunohistochemistry or Elisa method.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian L. Siu, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Razak AR, Hotte SJ, Siu LL, Chen EX, Hirte HW, Powers J, Walsh W, Stayner LA, Laughlin A, Novotny-Diermayr V, Zhu J, Eisenhauer EA. Phase I clinical, pharmacokinetic and pharmacodynamic study of SB939, an oral histone deacetylase (HDAC) inhibitor, in patients with advanced solid tumours. Br J Cancer. 2011 Mar 1;104(5):756-62. doi: 10.1038/bjc.2011.13. Epub 2011 Feb 1. PMID 21285985